CLINICAL TRIAL: NCT05821543
Title: An Open-label, Multicentre, Randomized Comparative Study to Evaluate the Efficacy and Safety of Using the Sibutramin-containing Drugs Reduxin® Forte and Reduxin® in Patients With Alimentary Obesity
Brief Title: Efficacy and Safety of Sibutramin-containing Drugs in Patient With Alimentary Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI/0619-1
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Obesity
Keywords: obesity; sibutramine; metformin; Reduxin; Reduxin Forte; pharmacotherapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduxin Forte (Experimental): Arm 1 (n=120) received metformin+sibutramine p. o., 1 tablet (850 mg + 10 mg) once per day. On day 30 ± 1, in the absence of a 2 kg weight loss compared to the first visit, the dose was increased in accordance with the medical instruction. The therapy period was 180 days.
  Interventions: Drug: metformin+sibutramine
- Reduxin (Active Comparator): Arm 2 (n=120) received sibutramine+ microcrystalline cellulose (MCC) p. o., 1 capsule (10 mg + 158.5 mg) once per day in the morning. On day 30 ± 1, in the absence of a 2 kg weight loss compared to the first visit, the dose was increased in accordance with the medical instruction. The therapy period was 180 days.
  Interventions: Drug: sibutramine+ microcrystalline cellulose

INTERVENTIONS:
Drug: metformin+sibutramine — 1 tablet (850 mg + 10 mg) once per day in the morning, without chewing and followed with a glass of water, during meals, for 180 days. At Visit 3 (Day 30 ± 1), in the absence of a 2 kg weight loss compared to Visit1 (Day 1), the zero dose was increased to 1 tablet (850 mg + 15 mg)
  Other Names: Reduxin® Forte
  Arms: Reduxin Forte
Drug: sibutramine+ microcrystalline cellulose — 1 capsule (10 mg + 158.5 mg) once per day in the morning, without chewing and followed with a glass of water, during meals for, 180 days.At Visit 3 (Day 30 ± 1), in the absence of a 2 kg weight loss compared to Visit 1 (Day 1), the zero dose was increased to 1 capsule (15 mg + 153,5 mg)
  Other Names: Reduxin®
  Arms: Reduxin

SUMMARY:
This is Open multicenter randomized Phase IV study to evaluate the efficacy and safety of the drug Reduxin® Forte, film-coated tablets, in comparison with the drug Reduxin®, capsules, in patients with alimentary obesity was conducted in 5 cities of the Russian Federation (St. Petersburg, Ivanovo, Kirov, Samara, Rostov-on-Don) on the basis of 8 research centers.

DETAILED DESCRIPTION:
Male and female patients (240 people) inclusive with alimentary obesity, meeting the inclusion criteria and not meeting the non-inclusion criteria, were randomized into 2 groups in a 1:1 ratio. One group (n=120) received sibutramine+ metformin p. o., 1 tablet (850 mg + 10 mg) once per day, the second group (n=120) received sibutramine+ microcrystalline cellulose (MCC) p. o., 1 capsule (10 mg + 158.5 mg) once per day in the morning. On day 30 ± 1, in the absence of a 2 kg weight loss compared to the first visit, the dose was increased in accordance with the medical instruction. The therapy period was 180 days.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of the Informed Consent Form of the Patient Information Leaflet (PIL) signed and dated by patient.
2. Men and women aged 18 to 65 years inclusive at the time of signing the Informed Consent Form in PIL.
3. The presence of alimentary obesity.
4. BMI >30 kg/m2.
5. Failure of non-pharmacological treatment at the time of screening (weight loss <5% within 3 months of treatment).
6. Patient consent to change in diet, eating behavior, and increased physical activity, and adherence to the investigator's recommendations throughout participation in the study
7. Patient's consent to use reliable contraceptive methods through out the study and for 3 weeks after the end of the study. The following people could take part in the study:

   * women who have a negative pregnancy test and use the following contraceptive methods: a barrier method (condom or occlusive cap (diaphragm or cervical/vaulted cap)) or a double barrier method of contraception (condom or occlusive cap). The use of estrogen-containing contraceptives was allowed provided that the drug was used in one dosing regimen for at least 3 months prior to study entry and it was planned to use it at the same dosing regimen throughout the study participation. Women incapable of childbearing may also participate in the study (with past history of: hysterectomy, tubal ligation, infertility, menopause for more than 1 year) or
   * men with preserved reproductive function using barrier contraceptives, as well as men with infertility or a history of vasectomy

Exclusion Criteria:

1. Hypersensitivity to the components of the study drug/comparator drug
2. Secondary (symptomatic) obesity.
3. Diabetes mellitus type I or II in history and/or at the time of screening.
4. Use of a low-calorie (<1600 kcal/day) diet for 3 months prior to screening.
5. Patients who previously received drugs based on sibutramine.
6. The use of drugs, herbal remedies or dietary supplements for the treatment of obesity less than 3 months prior to screening.
7. Use of systemic glucocorticosteroids for less than 3 months prior to screening.
8. Plan to change current smoking status during the study or quit smoking less than 3 months prior to screening.
9. The need for surgical treatment of obesity during the study or the history of this treatment.
10. Impaired liver function (AST and/or ALT ≥ 2 UNL and/or total bilirubin ≥ 1.5 UNL) at the time of screening.
11. Impaired renal function (creatinine clearance, calculated according to the Cockcroft- Gault formula, less than 45 ml/min) at the time of screening.
12. Acute conditions in which there was a risk of developing impaired renal function:

    dehydration (with diarrhea, vomiting), severe infectious diseases, shock (at the time of screening).
13. Cardiovascular diseases (in history and/or at the time of screening): ischemic heart disease (myocardial infarction, angina pectoris), chronic heart failure in the stage of decompensation, occlusive diseases of peripheral arteries, tachycardia (HR> 90 beats/min (mean for 3 measurements)), arrhythmia, cerebrovascular diseases (stroke, transient disorders of cerebral circulation).
14. Uncontrollable hypertension (blood pressure (BP) >145/90 mm Hg on screening).
15. History of pulmonary hypertension.
16. Clinically apparent manifestations of acute and chronic diseases that could lead to the development of tissue hypoxia (including respiratory failure, heart failure).
17. Hyperthyroidism.
18. Uncontrolled hypothyroidism at the time of screening (if using thyroid drugs or synthetic thyroid hormones, the drugs must have been used at a stable dose for at least 3 months prior to screening).
19. Subclinical hypothyroidism at the time of screening.
20. Benign prostatic hyperplasia (for men) in history.
21. Pheochromocytoma in history or suspicion of its presence at screening.
22. Angle-closure glaucoma in history.
23. Lactic acidosis (in history and at the time of screening).
24. Chronic alcoholism, acute ethanol poisoning at the time of screening.
25. Pharmacological and drug dependence in history and / or at the time of screening.
26. Serious eating disorders (anorexia nervosa, bulimia nervosa).
27. History of cholelithiasis or presence of symptoms of cholelithiasis within 3 months prior to screening.
28. History of schizophrenia, schizoaffective disorder, bipolar disorder, or other psychiatric disorder or suspected of having them at the time of screening.
29. History of suicide attempt.
30. Syndrome of Gilles de la Tourette (generalized tics) in history.
31. Major surgery or trauma (associated with a risk to the patient's life) in the last 6 months before screening.
32. Planned surgery (elective surgery) at the time of screening
33. Uncontrolled asthma or asthma controlled by steroids.
34. History of seizures (with the exception of febrile seizures in childhood) or an increased risk of developing seizures.
35. HIV, viral hepatitis B and/or C, history of active tuberculosis.
36. The need for the use of drugs from the list of prohibited therapies.
37. Taking other medications that, in the opinion of the investigator, could affect the course and results of the clinical trial.
38. History of malignant neoplasms, except for patients who have not been observed for the disease within the last 5 years, patients with completely healed basal cell skin cancer or completely healed carcinoma in situ.
39. Severe, decompensated or unstable somatic diseases (any disease or condition that threatened the patient's life or worsened the patient's prognosis, and also made it impossible for him to participate in a clinical study).
40. Patient's unwillingness or inability to comply with procedures of the Study Protocol (in the opinion of the investigator).
41. Pregnancy or breastfeeding period (for women).
42. Participation in another clinical trial within 3 months prior to study enrollment.
43. Other conditions that, in the opinion of the investigator, prevented the inclusion of the patient in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
The rate of achieving >5% weight loss | From baseline to Visit 13 (study completion, 180 days)
  The proportion of patients who had achieved more than 5% weight loss

SECONDARY OUTCOMES:
The frequency of patients who required an increase in the dose of the study / reference drug | From baseline to Visit 3 (30±1 days)
  The proportion of the patients requiring an increase in the study / reference dose
The magnitude of the change in body weight | From baseline to Visit 13 (study completion, 180 days)
  Value of weight change calculated as weight on Visit 13 to baseline (kg)
The change in Body Mass Index (BMI) | From baseline to Visit 13 (study completion, 180 days)
  The average value of the change in BMI (%)
The dynamic of body weight | From baseline to Visit 13 (study completion, 180 days)
  The mean body weight by each two weeks (kg)
The dynamic of BMI | From baseline to Visit 13 (study completion, 180 days)
  The average value of BMI by every month (kg/m2)
The dynamic of waist measurement | From baseline to Visit 13 (study completion, 180 days)
  The average waist measurement by every month(cm)
The dynamic of hip width | From baseline to Visit 13 (study completion, 180 days)
  The average hip width by every month(cm)
The dynamic of waist / hip measurements | From baseline to Visit 13 (study completion, 180 days)
  The average value of the ratio waist / hip measurements by every month
Dynamics of lipid profile indicators (TG, total cholesterol, LDL-cholesterol, HDL-cholesterol) | From baseline to Visit 13 (study completion, 180 days)
  The mean value of triglyceride, total cholesterol, LDL- cholesterol, HDL - cholesterol (mmol/l) by every month
The dynamic of quality of life | From baseline to Visit 13 (study completion, 180 days)
  The data obtained using the SF-36 Quality of life questionnaire, the average score of the physical health and psychological health by every month

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Demidova, Principal Investigator — Pirogov Russian National Research Medical University
Locations (8):
- Russia (8):
  - Ivanovo Clinical Hospital named after Kuvaev, Ivanovo
  - Kirov State Medical University, Kirov
  - Pirogov Russian National Research Medical University, Moscow
  - "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don
  - "Clinical hospital "RZD-Medicine" of the city of St. Petersburg", Saint Petersburg
  - Avrora Limited Liability Company Principal, Saint Petersburg
  - Limited Liability Company "Medica", Saint Petersburg
  - OrKli Hospital Limited Liability Company, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Demidova T.Yu., Izmailova M.Y., Ushakova S.E., Zaslavskaya K.Y., Odegova A.A., Popova V.V., Nevretdinova M.E., Bely P.A. EVALUATION OF WEIGHT REDUCTION EFFICACY AND SAFETY OF SIBUTRAMIN-CONTAINING DRUGS IN PATIENTS WITH ALIMENTARY OBESITY. Pharmacy & Pharmacology. 2022;10(3):289-304. https://doi.org/10.19163/2307-9266-2022-10-3-289-304
- See also: "Pharmacy & Pharmacology" ("Farmatsiya i farmakologiya") peer-reviewed scientific Journal is meant for scintifical and educational pharmaceutical and medical establishments, pharmaceutical enterprises, research organizations. — http://www.pharmpharm.ru/jour/article/view/1121